CLINICAL TRIAL: NCT06651476
Title: A Randomized Controlled Trial to Test Whether Oxytocin Amplifies the Effect of Vibration to Increase Heat Pain Threshold After UV-B Burn
Brief Title: A Randomized Controlled Trial to Test the Effects Oxytocin and Vibration Have on Heat Pain Threshold After UV-B Burn
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB00120861; 5P01NS119159 (NIH)
Record Dates: First submitted 2024-10-17; First posted 2024-10-21 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-11

CONDITIONS: Sunburn
Keywords: healthy volunteer; UVB burn; burn pain
MeSH Terms: conditions — Sunburn; Pain | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- oxytocin (Experimental): Two 30 minute infusions of oxytocin, 10 International Units (IU) separated by 30 minutes. To avoid potential unmasking by facial flushing which can occur at the beginning of high rates of oxytocin administration, the first infusion will consist of two steps beginning with a rate of 0.125 IU oxytocin per minute for 5 minutes, then increased to 0.375 IU oxytocin for 25 minutes. The second infusion will be a constant rate of 0.333 IU oxytocin per minute for 30 minutes.
  Interventions: Drug: oxytocin
- placebo (Placebo Comparator): Two 30 minute infusions of placebo separated by 30 minutes. The first infusion will consist of two steps, using an equivalent volume of placebo fluid infusion as in the oxytocin arm. This will consist of a slower rate in the first 5 minutes and more rapid rate for the last 25 min. The second placebo solution infusion will be a constant rate and volume equivalent to that used in the oxytocin arm.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: oxytocin — Oxytocin 10 IU will be administered over 30 minutes by intravenous infusion and repeated 30 minutes after the end of the first infusion.
  Arms: oxytocin
Drug: placebo — A placebo will be administered over 30 minutes by intravenous infusion and repeated 30 minutes after the end of the first infusion.
  Arms: placebo

SUMMARY:
This study aims to answer the question: Does oxytocin increase the pain threshold on thermal heat pain in the presence of vibration on an area of skin exposed to a mild sunburn?

DETAILED DESCRIPTION:
The goal of this clinical trial is to test whether intravenous oxytocin increases the analgesic effect of vibration on heat pain threshold of skin that has been exposed to Ultraviolet-B (UV-B) burn (mild sunburn). Researchers will compare oxytocin (a hormone that naturally occurs in the body) to a placebo (a look-alike substance that contains no drug) to see if oxytocin works to increase the pain threshold (the lowest intensity at which one begins to perceive or sense a stimulus as being painful).

ELIGIBILITY:
Inclusion Criteria:

* Male or female > 18 and ≤55 years of age, Body Mass Index (BMI) <40
* Generally in good health as determined by the Principal Investigator based on prior medical history, and as assessed to be American Society of Anesthesiologists physical status 1, 2, or 3
* Fitzpatrick Scale rating I through III

Exclusion Criteria:

* History of skin cancer
* Dark enough skin complexion that would make it infeasible to determine the minimal erythematous dose of UV-B irradiation. Anyone Fitzpatrick Scale score >3 will be excluded
* Neuropathy, chronic pain (located in any body location that is being treated), diabetes mellitus, or taking benzodiazepines or pain medications on a daily basis
* Pregnancy or currently breast feeding
* Subjects with current or history of ventricular tachycardia, atrial fibrillation or prolonged QT interval
* Subjects with past or current history of hyponatremia or at risk for hyponatremia; anyone taking thiazide diuretics, loop diuretics, combination diuretics, lithium, carbamazepine, enalapril, Ramipril, celecoxib, temazepam, gliclazide, glimepiride, glibenclamide, glipizide, omeprazole, pantoprazole, desmopressin, SSRI's, MAOI, or the recreational drug ecstasy
* Subjects with a known latex allergy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2024-12-05 (Actual); Primary Completion 2025-11-20 (Actual); Study Completion 2025-11-20 (Actual)

PRIMARY OUTCOMES:
Difference between heat pain threshold | 24 hours after UV-B exposure
  Difference between heat pain threshold at 24 hours after Ultraviolet-B (UV-B) exposure at 3x minimum erythematous dose. The difference between the average threshold for stimuli #5-8 and the average threshold for stimuli #13-17 at baseline and 2 hours after the beginning of the oxytocin or placebo infusion will be used. The values are measured in degrees Celsius. A lower temperature indicates more sensitivity to heat pain.

SECONDARY OUTCOMES:
Difference between heat pain threshold | Two days after UV-B exposure
  Difference between heat pain threshold at 24 hours after UV-B exposure at 3x minimum erythematous dose. The difference between the average threshold for stimuli #5-8 and the average threshold for stimuli #13-17 at baseline and 2 days after the beginning of the oxytocin or placebo infusion will be used. The values are measured in degrees Celsius. A lower temperature indicates more sensitivity to heat pain.
Touch and pain threshold to von Frey filament application | 24 hours after UV-B exposure
  Using an electronic von Frey instrument, threshold for touch and a prickly pain sensation will be determined at the site of UV-B exposure at 3x minimum erythematous dose and in normal skin to estimate the threshold for touch and prickly pain sensation. The measure will be recorded in grams. A lower pressure indicates more sensitivity to touch and pain.
Touch and pain threshold to von Frey filament application | Two days after UV-B exposure
  Using an electronic von Frey instrument, threshold for touch and a prickly pain sensation will be determined at the site of UV-B exposure at 3x minimum erythematous dose and in normal skin to estimate the threshold for touch and prickly pain sensation. The measure will be recorded in grams. A lower pressure indicates more sensitivity to touch and pain.

CONTACTS AND LOCATIONS:
Overall Officials: James C Eisenach, M.D., Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Atrium Health Wake Forest Baptist Medical Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-10-08): https://cdn.clinicaltrials.gov/large-docs/76/NCT06651476/ICF_000.pdf